CLINICAL TRIAL: NCT03378011
Title: The Role of Long Wavelength UVA1 Phototherapy in Acral Vitiligo
Brief Title: UVA1 Phototherapy in Acral Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dermatology 3
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Acral Vitiligo
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UVA1 phototherapy (Active Comparator): UVA1 phototherapy in acral vitiligo
  Interventions: Other: phototherapy
- Topical PUVA (Active Comparator): Topical PUVA in acral vitiligo
  Interventions: Other: phototherapy

INTERVENTIONS:
Other: phototherapy — phototherapy either UVA1 or topical PUVA on acral vitiligo

SUMMARY:
evaluate the effect of UVA1 phototherapy in the treatment of acral vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acral vitiligo.
* Patients more than 12 years old.

Exclusion Criteria:

* Patients less than 12 years old.
* Patients with any other skin diseases or autoimmune diseases.
* Patients taking medical treatment or phototherapy for vitiligo.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
effect of medium dose UVA1 phototherapy in treatment of acral vitiligo | 1 year
  effect of medium dose UVA1 phototherapy in treatment of acral vitiligo using point counting and vitiligo area severity index (VASI) score

CONTACTS AND LOCATIONS:
Overall Officials: Maha Elmasry, Principal Investigator — Cairo University
Locations (1):
- Maha Fathy Elmasry, Cairo, Egypt